CLINICAL TRIAL: NCT03905265
Title: A Phase II, Randomized, Double-blind, Parallel Group Dose Finding Study of Single Oral Doses of Moxidectin in Adults With Scabies
Brief Title: Dose-finding Study of Moxidectin for Treatment of Scabies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medicines Development for Global Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDGH-MOX-2001
Record Dates: First submitted 2019-03-18; First posted 2019-04-05 (Actual); Results first posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2022-05

CONDITIONS: Scabies
Keywords: moxidectin; acaricide; oral
MeSH Terms: conditions — Scabies

STUDY DESIGN:
Intervention Model Description: Parallel, double blind, multicenter, randomized, pharmacokinetic/pharmacodynamic study. Three cohorts of six subjects per cohort are planned. Subjects will be randomized 1:1:1 to receive 2, 8 or 20 mg moxidectin as a single oral dose. An additional cohort of 36 mg may be initiated with a target sample size of 6 subjects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To maintain blinding to treatment allocation, all subjects will receive treatment with the same number of tablets, comprised of moxidectin 2 mg tablets and matched placebo (as required).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Moxidectin 2 mg (Experimental): Moxidectin 2 mg will be administered as a single dose. Each subject will receive the same number of tablets made up of moxidectin 2 mg tablets and placebo tablets to maintain the blind.
  Interventions: Drug: Moxidectin Oral Product
- Moxidectin 8 mg (Experimental): Moxidectin 8 mg will be administered as a single dose. Each subject will receive the same number of tablets made up of moxidectin 2 mg tablets and placebo tablets to maintain the blind.
  Interventions: Drug: Moxidectin Oral Product
- Moxidectin 20 mg (Experimental): Moxidectin 20 mg will be administered as a single dose. Each subject will receive the same number of tablets made up of moxidectin 2 mg tablets and placebo tablets to maintain the blind.
  Interventions: Drug: Moxidectin Oral Product
- Moxidectin 36 mg (Experimental): Moxidectin 36 mg will be administered as a single dose. Each subject will receive the same number of tablets made up of moxidectin 2 mg tablets and placebo tablets to maintain the blind.
  Interventions: Drug: Moxidectin Oral Product

INTERVENTIONS:
Drug: Moxidectin Oral Product — The required number of moxidectin 2 mg oral tablets will be administered as a single dose with placebo to match as required

SUMMARY:
The effective dose of moxidectin to treat human scabies is not known. This study aims to provide proof of concept that a single dose of moxidectin is effective in eliminating the scabies parasite in humans and to enable the determination of an optimal dose of moxidectin for treatment of scabies for further clinical studies.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years.
2. Provision of written informed consent.
3. Parasitologically confirmed active Sarcoptes scabiei infestation, defined as the presence of at least two lesions (which may include burrows), each containing at least one live (internal and/or external structures discernable) adult Sarcoptes scabiei mite observed by reflectance confocal microscopy.
4. Agree to the use of reliable contraceptive measures if female or male partner of a female of child-bearing potential from Screening and until 6 months after treatment with study product.

Exclusion Criteria:

1. History of chronic or recurring dermatologic disease (other than scabies) that could interfere with the diagnosis and/or subsequent clinical assessment of scabies.
2. Diagnosis of crusted/Norwegian scabies or scabies that, in the opinion of the Investigator, would require treatment with more than one standard of care (e.g. scabies requiring concurrent topical and oral treatment).
3. Received any treatment for scabies within 7 days of Screening, including but not limited to permethrin, ivermectin, benzyl benzoate, lindane, crotamiton, malathion, and/or tea tree oil.
4. Presence of any other clinically relevant condition, including infection, immunological disorder, malignant disease, and/or other underlying condition or circumstance at Screening or Baseline that would put the subject at increased risk from participating in the study or confound study evaluations.
5. Poor venous access.
6. Received an investigational agent within 28 days of Screening (or 5 half-lives of the investigational agent, whichever is longer).
7. Body Mass Index over 35 kg/m2.
8. Clinically relevant abnormal findings in vital signs, 12-lead electrocardiogram (ECG), or physical examination at Screening and/or Baseline in the opinion of the Investigator.
9. Clinically relevant laboratory abnormalities at Screening, including:

   1. alanine aminotransferase or aspartate aminotransferase > 2.5 x upper limit of reference range;
   2. creatinine > 2.0 milligrams per deciliter (mg/dL);
   3. hemoglobin < 9.5 g/dL (female) or <10.5 g/dL (male);
   4. amylase > 2.0 x upper limit of reference range.
10. Known or suspected hypersensitivity to macrocyclic lactones or excipients used in the formulation of moxidectin.
11. Use of systemic steroids within 14 days of Screening, or history of prolonged use of systemic and/or high-dose inhaled corticosteroids, or use of topical steroids for 7 out of the 14 days prior to Screening.
12. Subjects with known or suspected Loa loa coinfection.
13. Difficulty swallowing tablets.
14. Pregnant or breastfeeding, or planning to become pregnant.
15. Known or suspected alcohol or illicit substance abuse.
16. Unwilling, unlikely or unable to comply with all protocol specified assessments.
17. Previous enrolment and treatment with moxidectin in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Royal Darwin Hospital, Darwin, Australia
- Medizinischen Universität Wien, Vienna, Austria
- France (3):
  - Hopital Henri Mondor AP-HP, Créteil
  - CHU Nice Hopital Archet 2, Nice
  - CHU Saint-Etienne Hopital Nord, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was open to recruitment on 13 Jan 2020 and the First participant was screened on 15 Jan 2020. Last participant last study visit was completed on 28 Feb 2022.
Groups:
- Moxidectin 2 mg: 4 Participants received Moxidectin 2 mg as a single dose. Each participant received the same number of tablets made up of moxidectin 2 mg tablets and placebo tablets to maintain the blind.
  Moxidectin Oral Product: 2 mg oral tablets
- Moxidectin 8 mg: 4 Participants received Moxidectin 8 mg as a single dose. Each participant received the same number of tablets made up of moxidectin 2 mg tablets and placebo tablets to maintain the blind.
  Moxidectin Oral Product: 8 mg oral tablets
- Moxidectin 20 mg: 6 Participants received Moxidectin 20 mg as a single dose. Each participant received the same number of tablets made up of moxidectin 2 mg tablets and placebo tablets to maintain the blind.
  Moxidectin Oral Product: 20 mg oral tablets
- Moxidectin 36 mg: 8 Participants received Moxidectin 36 mg as a single dose.
  Moxidectin Oral Product: 36 mg oral tablets
Period: Overall Study
Arm/Group | Moxidectin 2 mg | Moxidectin 8 mg | Moxidectin 20 mg | Moxidectin 36 mg
Started | 4 | 4 | 6 | 8
Completed | 3 (1 participant withdrew from study prematurely due to withdrawal of consent.) | 3 (1 participant withdrew from study prematurely due to withdrawal of consent.) | 6 | 8
Not Completed | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis Population is all enrolled subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Moxidectin 2 mg | Moxidectin 8 mg | Moxidectin 20 mg | Moxidectin 36 mg | Total
Number analyzed (Participants) | 4 | 4 | 6 | 8 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6 | 7 | 19
  >=65 years | 1 | 1 | 0 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (18.88) | 45.3 (15.50) | 27.2 (9.33) | 29.4 (17.26) | 34.8 (16.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 4 | 4 | 13
  Male | 0 | 3 | 2 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 2 | 3 | 4 | 8 | 17
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 2 | 0 | 5
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: One subject did not have height or weight measured at Baseline, therefore a BMI could not be derived for this subject hence n=3 for this parameter.
  kg/m^2
    number analyzed (Participants) | 4 | 3 | 6 | 8 | 21
    (all) | 32.98 (9.95) | 25.27 (2.40) | 21.70 (2.31) | 28.68 (8.46) | 27.01 (7.68)

OUTCOME MEASURES:

1. Primary Outcome: Mortality Rate for Adult Scabies Mites
Description: Adult scabies mite death was based on the reflectance confocal microscopy (RCM) morphology assessment of 2 live adult scabies mites nominated pre-treatment (Baseline), hence overall number of units analyzed are different from the overall number of participants. For the outcome measure, the number of adult mites assessed at each timepoint is the sum of the number of adult mites from all participants in the analysis population for each dose. Therefore, mortality was assessed in 2 mites in the 2 mg group, 6 in the 8 mg group, 8 in the 20 mg group and 14 in the 32 mg group. Adult mite death was defined as the degradation (homogenization of internal structures and/or external anatomic structures, and increased reflectance) of the adult mite observed by RCM. The number of dead mites was assessed at Hours 4, 8, 24, 48 and 72, and Days 7, 14 and 28 compared to the baseline adult mites.
Time Frame: 28 days
Population: Per protocol analysis set
Measure: Number; unit: Adult mites
Units Other Than Participants: Total number of live adult mites
Arm/Group | Moxidectin 2 mg | Moxidectin 8 mg | Moxidectin 20 mg | Moxidectin 36 mg
Number analyzed (Participants) | 1 | 3 | 4 | 7
Number analyzed (Total number of live adult mites) | 2 | 6 | 8 | 14
Adult mites
  Number of live adult mites assessed at Baseline | 2 | 6 | 8 | 14
  Number of dead adult mites assessed at Day 0-4 hours timepoint | 0 | 0 | 0 | 0
  Number of dead adult mites assessed at Day 0-8 hours timepoint | 0 | 1 | 0 | 0
  Number of dead adult mites assessed at Day 1 timepoint | 0 | 2 | 0 | 0
  Number of dead adult mites assessed at Day 2 timepoint | 0 | 2 | 1 | 2
  Number of dead adult mites assessed at Day 3 timepoint | 0 | 2 | 2 | 3
  Number of dead adult mites assessed at Day 7 timepoint | 0 | 4 | 4 | 9
  Number of dead adult mites assessed at Day 14 timepoint | 0 | 5 | 8 | 12
  Number of dead adult mites assessed at Day 28 timepoint | 0 | 6 | 8 | 14

2. Primary Outcome: Summary of Participants With Most Commonly Occurring Adverse Events by Preferred Term (Safety Analysis Set)
Description: No formal statistical analysis of AEs was undertaken. Adverse events reported in this Section refer to treatment emergent adverse events (TEAE), defined as AEs that started, or worsened, on or after the start of the administration of Investigational Product (Moxidectin). Moxidectin was generally well tolerated, with no treatment-related SAEs reported and no treatment emergent adverse event (TEAEs) leading to study withdrawal or resulting in death. Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term. Data up to and including the Day 28 assessment for each subject.
Time Frame: Day 0 to Day 28 inclusive
Population: The Safety Analysis Set (SfAS) included all subjects exposed to study drug. Subjects were analyzed according to the actual dose of study drug received regardless of their randomized dose group. Unless otherwise noted, the SfAS was used for all safety analyses. Reported data table represent the number of participants with most commonly occurring Adverse Events by Preferred Term.
Measure: Count of Participants; unit: Participants
Arm/Group | Moxidectin 2 mg | Moxidectin 8 mg | Moxidectin 20 mg | Moxidectin 36 mg
Number analyzed (Participants) | 4 | 4 | 6 | 8
Participants
  Infections and infestations | 3 | 3 | 5 | 5
  Skin and subcutaneous tissue disorder | 1 | 2 | 1 | 4
  Nervous system disorders | 2 | 0 | 1 | 3
  Psychiatric disorders | 2 | 0 | 1 | 0
  Gastrointestinal disorders | 0 | 1 | 1 | 0

3. Primary Outcome: Number of Participants and Severity of Adverse Events
Description: Number of participants with Adverse events reported in this Section refer to treatment emergent adverse events (TEAE), defined as AEs that started, or worsened, on or after the start of the administration of IP. Data up to and including the Day 28 assessment for each subject. The severity of adverse events were assessed using the Toxicity Grading Scale for Healthy Adult and Adolescent volunteers Enrolled in Preventive Vaccine Clinical Trials.
Time Frame: Day 0 to Day 28 inclusive
Population: The Safety Analysis Set (SAS) included all subjects exposed to study drug. Subjects were analyzed according to the actual dose of study drug received regardless of their randomized dose group. Unless otherwise noted, the SfAS was used for all safety analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Moxidectin 2 mg | Moxidectin 8 mg | Moxidectin 20 mg | Moxidectin 36 mg
Number analyzed (Participants) | 4 | 4 | 6 | 8
Participants
  Grade 1 TEAEs | 1 | 1 | 4 | 5
  Grade 2 TEAEs | 3 | 3 | 2 | 3
  Grade 3 TEAEs | 0 | 0 | 0 | 0
  Grade 4 TEAEs | 0 | 0 | 0 | 0

4. Secondary Outcome: Analysis of Moxidectin Plasma Concentrations
Description: The final PK analysis dataset included a total of 240 evaluable PK samples from 22 subjects. All pre-dose samples were below the limit of quantitation (BQL).
Time Frame: Nominal time of PK sample collection was Pre-dose, 2hours (h), 3h, 4h, 8h, Day 1 (24h), Day 2 (48h), Day 3 (72h), Day 7 (168h), Day 14 (336h) and Day 28 (672h)
Population: Pharmacokinetic parameters were calculated and derived using non-compartmental methods. AUC calculation method was linear up log down.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Moxidectin 2 mg | Moxidectin 8 mg | Moxidectin 20 mg | Moxidectin 36 mg
Number analyzed (Participants) | 4 | 4 | 6 | 8
hr*ng/mL
  AUC0-24 (hr*ng/mL) | 181 (43.2) | 744 (37.9) | 1670 (40.2) | 2930 (26.8)
  AUC0-48 (hr*ng/mL) | 212 (44.2) | 903 (35.0) | 2000 (40.7) | 3560 (29.3)
  AUC0-72 (hr*ng/mL) | 229 (45.5) | 989 (33.7) | 2200 (40.4) | 3900 (31.0)
  AUC0-D7 (hr*ng/mL) | 276 (50.6) | 1230 (30.5) | 2780 (39.5) | 4770 (35.1)
  AUC0-D14 (hr*ng/mL) | 329 (62.8) | 1540 (27.9) | 3530 (39.3) | 5820 (38.1)
  AUC0-D28 (hr*ng/mL) | 408 (82.5) | 1970 (30.0) | 4670 (41.1) | 7430 (37.6)

5. Secondary Outcome: Analysis of Moxidectin Maximum Plasma Concentrations (Cmax)
Description: as for outcome 4
Time Frame: as for outcome 4
Population: Cmax was calculated and derived using non-compartmental methods.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Cmax (ng/mL)
Arm/Group | Moxidectin 2 mg | Moxidectin 8 mg | Moxidectin 20 mg | Moxidectin 36 mg
Number analyzed (Participants) | 4 | 4 | 6 | 8
Cmax (ng/mL) | 21.0 (47.1) | 73.5 (42.0) | 207 (44.9) | 277 (26.9)

6. Other Pre Specified Outcome: Incidence and Severity of Scabies Signs and Symptoms
Description: The incidence and severity of signs and symptoms of scabies infection will be explored using a clinician-reported scabies severity assessment.
Time Frame: 28 days
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Severity of Pruritus
Description: The severity of pruritus will be determined using the Numerical Rating Scale where 0="no itch" and 10="worst itch imaginable"
Time Frame: 28 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Day 0 to Week 12, inclusive.
Description: Treatment-emergent adverse events (TEAEs) were defined as adverse events that started or worsened on or after the start of investigational product administration. TEAEs that occurred in more than 5% of subjects overall are reported. The most commonly occurring TEAEs are defined as those occurring in two or more subjects (5%) overall.
Arm/Group | Moxidectin 2 mg | Moxidectin 8 mg | Moxidectin 20 mg | Moxidectin 36 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/6 | 1/8
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 6/6 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moxidectin 2 mg (N=4) | Moxidectin 8 mg (N=4) | Moxidectin 20 mg (N=6) | Moxidectin 36 mg (N=8)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moxidectin 2 mg (N=4) | Moxidectin 8 mg (N=4) | Moxidectin 20 mg (N=6) | Moxidectin 36 mg (N=8)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 2 (2) | 3 (3) | 4 (5) | 5 (6)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Small number of subjects, especially in the per-protocol analysis set, confounds interpretation of some study results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution agrees that no Publication of the Study results may be made until Publication of the results of the Study or 2 years after Study Completion, whichever is the sooner.

The Institution must ensure that the Discloser gives a copy of any proposed Publication drafted by them and/or other Personnel involved in the conduct of the Study to the Sponsor at least 40 days before forwarding it to any person that is not bound by the confidentiality obligations

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/65/NCT03905265/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/65/NCT03905265/SAP_001.pdf